CLINICAL TRIAL: NCT01598623
Title: A Randomized Trial Administering Oxytocin vs Placebo as add-on to Antipsychotics in Patients With Schizophrenia and Schizo-affective Disorder
Brief Title: Administrating Oxytocin to Treat Treatment Schizophrenia and Schizo-affective Patients
Acronym: OXY-S-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-12-9103-MW-CTIL
Record Dates: First submitted 2012-05-03; First posted 2012-05-15 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Oxytocin + Non Specific Counselling; Oxytocin + Social Skills Training; Placebo + Non Specific Counselling; Placebo + Social Skills Training
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oxytocin+ Non Specific Counselling (Experimental)
  Interventions: Drug: Oxytocin
- Oxytocin + Social Skills training (Experimental)
  Interventions: Drug: Oxytocin; Behavioral: Social Skills Training
- Placebo + Non Specific Counselling (Placebo Comparator)
  Interventions: Behavioral: Placebo + Non Specific Counselling
- Placebo + Social Skills Training (Experimental)
  Interventions: Behavioral: Social Skills Training

INTERVENTIONS:
Drug: Oxytocin — 24 IU Intranasal, three times daily (morning, noon and evening, before meals) for 3 weeks (21 days).
  Arms: Oxytocin + Social Skills training; Oxytocin+ Non Specific Counselling
Behavioral: Social Skills Training — three times a week for three weeks.
  Arms: Oxytocin + Social Skills training; Placebo + Social Skills Training
Behavioral: Placebo + Non Specific Counselling
  Arms: Placebo + Non Specific Counselling

SUMMARY:
The objectives of the study are:

1. To evaluate the effect of OT compared to placebo, as add-on to anti-psychotics, on social functioning in schizophrenia.
2. To evaluate the effect of socially oriented CBT administered to patients immediately after they receive OT, compared to patients who receive OT with not-socially oriented CBT, and compared to patients who receive socially oriented CBT without OT. The investigators hypothesize that OT and socially oriented CBT will have a synergistic effect, and will be better than OT or CBT alone.
3. Use a detailed, in depth analysis of social interaction to assess these putative effects of OT. The investigators hypothesize that the use of this analysis will show larger treatment effects of OT than previously shown in less sensitive assessments, such as PANSS.
4. To assess the effect of epigenetic status on response to OT. The investigators hypothesize that epigenetic variants associated with lower OT plasma levels will be associated with greater response to OT treatment.
5. To assess in the relationships between levels of salivary OT and vasopressin, and social interactions in schizophrenia.
6. To assess in the relationships between levels of salivary OT and vasopressin, and response to OT treatment.

DETAILED DESCRIPTION:
Social disability is a hallmark of schizophrenia, and improving social functioning in schizophrenia should improve patients' overall functioning and quality of life. Oxytocin (Granholm, McQuaid et al.) is a nine amino-acid neuropeptide synthesized in the hypothalamus, has found to modulate social behaviors in mammals, including humans (Insel and Young 2001; Kosfeld, Heinrichs et al. 2005). Among its influences on human social behavior are increased trust (Kosfeld, Heinrichs et al. 2005), empathy (Hurlemann, Patin et al. 2010) and eye contact (Guastella, Mitchell et al. 2008).

Impaired social behaviors are a core domain of Autism Spectrum Disorders (ASD) (Modahl, Green et al. 1998; Bartz and Hollander 2008); studies have shown that social disabilities have been associated with OT dysfunction in ASD, and have been improved by administration of intranasal OT (Hollander, Bartz et al. 2007; Andari, Duhamel et al. 2010; Guastella, Einfeld et al. 2010).

Furthermore, epigenetic changes in the genes encoding for OT have been demonstrated in autism (Gregory, Connelly et al. 2009)

Impaired social functioning is a hallmark of schizophrenia; studies show that plasma levels of endogenous OT are lower in schizophrenia patients compared to controls, and patients with lower levels of plasma OT have more positive symptoms (Kéri , Kiss et al. 2009; Kיri, Kiss et al. 2009; Rubin, Carter et al. 2010). Moreover, a recent study demonstrated a significant genetic association between OT and Arginine Vasopressin, another peptide linked with social behavior, and schizophrenia (Teltsh, Kanyas-Sarner et al. 2011). Only two published studies have investigated the therapeutic potential of OT in schizophrenia; both administered OT in addition to anti-psychotic treatment. Feifel (Feifel, Macdonald et al. 2010) reported a decrease in positive symptoms after 3 weeks of treatment, and Pedersen (Pedersen, Gibson et al. 2011) reported an improvement in social cognition. There is ongoing research aiming to validate these findings.

Vasopressin is also a peptide with a putative effect on social interaction (Ebstein, Israel et al. 2009; Heinrichs, von Dawans et al. 2009). In this proposed study we will assay salivary levels both of OT and vasopressin.

In this proposed study we intend to administer OT in a placebo-controlled, double-blind design to patients with schizophrenia. In addition to assessing the effect of OT on the symptoms of schizophrenia, this proposal has four characteristics which we believe are unique, and we hope will enable a large step forward in understanding the role of OT in schizophrenia.

* Social functioning: will be assessed using previously validated techniques, by video-taping interviews with schizophrenia patients. The quality of the social interactions will then be assessed, by raters blinded to treatment status. The assessment will , specifically focus on the gaze to the experimenter's face, vocalization (patient's vocal output, positive/negative tone, and fluent speech) and affect, body tone, movements, and other non-verbal signs. This technique was developed in Prof. Feldman's lab, and has been show to accurately assess social interactions (Feldman, Masalha et al. 2001; Feldman and Klein 2003; Feldman and Eidelman 2009; Feldman 2010). This technique will enable meticulous quantification of the putative effects of OT on social functioning in schizophrenia.
* Data from preclinical models of traumatic brain injury (Feeney, Gonzalez et al. 1982) and clinical studies in stroke patients (Crisostomo, Duncan et al. 1988; Scheidtmann, Fries et al. 2001; Taub, Uswatte et al. 2002)] suggest that new learning develops faster, has increased magnitude and is longer lasting under a combined intervention of drug and practice relative to learning occurring under either intervention in isolation. Similar thoughts have been expressed regarding compounds which putatively enhance cognition, in that patients who receive compounds which enhance cognition should be treated with cognitive remediation at the same time. We propose to apply this concept to OT. In this proposal, patients will be treated with cognitive-behavioral therapy (socially oriented CBT) focused on social interactions, emphasizing eye contact, body language, empathy, etc. Socially oriented CBT will be administered three times/week during the time period immediately after OT administration, when OT is active. There will be a control CBT condition addressing medication compliance and vocational rehabilitation, without any social orientation, with somewhat analogous demand characteristics. We hypothesize that the combined effects of OT co-administered with socially oriented CBT will be synergistic, i.e. greater than the effect of either alone.
* The effects of epigenetic variation on the effects of OT treatment will be examined by assessing epigenetic status of subjects, and these will be correlated with response to treatment. We will examine the methylation status of two CpG sites (-934 and -924) in the OXTR promoter. The epigenetic evaluation would detect whether the exogenously administered OT changes OXTR genes, their expression or function on OT levels and behavior.
* Two previous studies have administered 40 international units (IU) X2/d= 80 IU/d (Feifel, Macdonald et al. 2010) or 24 IU X2/d= 48 IU/d (Pedersen, Gibson et al. 2011), with no adverse effects. Based on this data, we propose to administer 24 IU X3/d= 72 IU. This dose is lower than Feifel et al. and no adverse effects were seen. Therefore, we are sure that thus dose is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age, inclusive
2. Females who are abstinent or practicing an established method of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device [IUD]).
3. Willing and able to provide informed consent, after the nature of the study has been fully explained
4. Current DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder as confirmed by modified SCID.
5. Symptoms: PANSS total score ≤75
6. A score of 4 (moderate) or higher on at least one, or more of the following PANSS negative items: emotional withdrawal, poor rapport, passive-apathetic social withdrawal
7. Receiving the same antipsychotic medication for 2 weeks before randomization.
8. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission, provided no medication change since hospitalization.
9. Adjunctive treatment with anticholinergic agents, beta-blockers, mood stabilizers, antidepressants; and anxiolytics will be allowed provided that patients have been on the medication for at least 2 weeks prior to entry into the screening phase of the study.

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions.
2. Pregnant or breast-feeding.
3. Clinically significant medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning).
4. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
5. Patients with a current DSM-IV substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
6. Concurrent delirium, mental retardation, drug-induced psychosis, or history of clinically significant brain trauma documented by CT or MRI.
7. Patients with significantly impaired renal or liver function, defined as GOP and or GPT levels >3 times above highest normal value, and or blood creatinine levels above 1.5 will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-02 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Total score of structured assessment of social interaction | Baseline and week 3
  Change from baseline in the total score of structured assessment of social interaction in Oxytocin compared with placebo on all patients.

SECONDARY OUTCOMES:
Total score of structured assessment of social interaction | Total score of structured assessment of social interaction at week 3
  Change from baseline in the in Oxytocin with and without social skills training compared with placebo with and without social skills training.
PANSS positive, negative and general psychopathology scales scores | PANSS positive, negative and general psychopathology scales scores at week 1
  Change from baseline in Oxytocin compared with placebo on PANSS positive, negative and general psychopathology scales scores at 1 week
Total score of structured assessment of social interaction and PANSS scores, genetic and epigenetic status | Total score of structured assessment of social interaction and PANSS scores, genetic and epigenetic status at week 3
  Correlation between response to OT treatment(change from baseline in total score of structured assessment of social interaction and PANSS scores), genetic(types of variants of the OXT and OXTR genes)and epigenetic status(methylation on these genes) at 3 weeks
Levels of salivary OT,genetic,epigenetic status and total score of structured assessment of social interaction and PANSS scores. | Levels of salivary OT,genetic and epigenetic status at week 3
  Correlations between levels of salivary OT,genetic(type of variants of the OXT and OXTR genes),epigenetic(methylation on these genes)and response to OT treatment(change in total score of structured assessment of social interaction and PANSS scores) at 3 weeks
PANSS positive, negative and general psychopathology scales scores | PANSS positive, negative and general psychopathology scales scores at week 2
  Change from baseline in Oxytocin compared with placebo on PANSS positive, negative and general psychopathology scales scores at 2 weeks
PANSS positive, negative and general psychopathology scales scores | PANSS positive, negative and general psychopathology scales scores at week 3
  Change from baseline in Oxytocin compared with placebo on PANSS positive, negative and general psychopathology scales scores at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

REFERENCES:
- [Derived] Saporta-Wiesel L, Feldman R, Levi L, Davidson M, Burshtein S, Gur R, Zagoory-Sharon O, Amiaz R, Park J, Davis JM, Weiser M. Intranasal Oxytocin Combined With Social Skills Training for Schizophrenia: An Add-on Randomized Controlled Trial. Schizophr Bull Open. 2024 Oct 21;5(1):sgae022. doi: 10.1093/schizbullopen/sgae022. eCollection 2024 Jan. PMID 39502135